CLINICAL TRIAL: NCT02384304
Title: Guided and Unguided Internet Treatment for Problematic Alcohol Use: A Randomized Pilot Study
Brief Title: Guided and Unguided Internet Treatment for Problematic Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/1761-31/5
Record Dates: First submitted 2015-02-26; First posted 2015-03-10 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Alcohol Abuse; Alcohol Addiction
Keywords: randomized controlled trial; alcohol; internet; internet based therapy; cognitive behavior therapy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Choice (Experimental): A self help program consisting of 8 modules. Patients will have access to therapist support through either messages or chat sessions
  Interventions: Behavioral: Choice
- Messages (Experimental): A self help program consisting of 8 modules. Patients will have access to therapist support through messages
  Interventions: Behavioral: Messages
- Self help (Active Comparator): A relapse intervention program consisting of 8 modules. Patients will have no access to therapist support
  Interventions: Behavioral: Self help

INTERVENTIONS:
Behavioral: Choice — A self help program consisting of 8 modules and access to therapist guidance either through messages or through chat sessions
  Arms: Choice
Behavioral: Messages — A self help program consisting of 8 modules and access to therapist guidance through messages
  Arms: Messages
Behavioral: Self help — A self help program consisting of 8 modules
  Arms: Self help

SUMMARY:
The purpose of this study was to determine whether a 10-week internet-based program based on cognitive behavioral therapy (CBT) is effective in the treatment of alcohol problems, and if having therapist guidance leads to greater effects.

DETAILED DESCRIPTION:
Objectives: An 10 week Internet-based self-help program based on cognitive behavioral therapy (CBT) was tested among Internet help seekers.The design was a three-armed randomized controlled design, and outcomes were measured in terms of changes in problematic alcohol use, as well as depression, anxiety and quality of life. 80 participants were recruited entirely online from an open access website and randomized into three different groups. All participants had access to the same self-help program. However, one group was given a choice between two forms of therapist guidance (messages or weekly chat sessions), one group received therapist guidance in the form of secure messages, and one group received no therapist guidance.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* access to the Internet
* problematic alcohol use defined as ≥ 8 p or more for men and ≥ 6 p or more for women in the Alcohol Use Identification Scale

Exclusion Criteria:

• not adequately fluent in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back (TLFB) | Baseline and 10 weeks
  Change in total TLFB score (consumption during preceding week), as a summarized measure of alcohol consumption

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | Baseline and 10 weeks
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems)
Hamilton Anxiety and Depression Scale (HADS) | Baseline and 10 weeks
  Change in total HADS score, as a summarized measure of depression and anxiety, respectively
EQ5 | Baseline and 10 weeks
  Change in total EQ5 score, as a summarized measure of quality of life
WHOQOL-BREF | Baseline and 10 weeks
  Change in total WHOQOL-BREF score, as a summarized measure of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neuroscience, Center for Psychiatric Research, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Background] Sundström, C., Berman, A. H., Sinadinovic, K., & Johansson, M. (2013). Internet-based relapse prevention with therapist support for help-seeking problematic alcohol users: a randomized pilot study. Addiction science & clinical practice, 8(1), 1-1.
- [Derived] Sundstrom C, Gajecki M, Johansson M, Blankers M, Sinadinovic K, Stenlund-Gens E, Berman AH. Guided and Unguided Internet-Based Treatment for Problematic Alcohol Use - A Randomized Controlled Pilot Trial. PLoS One. 2016 Jul 6;11(7):e0157817. doi: 10.1371/journal.pone.0157817. eCollection 2016. PMID 27383389